CLINICAL TRIAL: NCT02085044
Title: Non Randomized Controlled Intervention Study Comparing Two Interventions of Nutritional Supplement on Malnutrition, Health and Mortality in Children Aged 6 to 24 Month Hadjer-Lamis Region - Chad
Brief Title: Non Randomized Controlled Intervention Study Comparing Two Interventions of Nutritional Supplement on Malnutrition, Health and Mortality
Acronym: NRCI-ASPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: France Broillet (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor-Investigator, France Broillet, Chargé de recherche operationnelle, Médecins Sans Frontières, Switzerland
Organization: Médecins Sans Frontières, Switzerland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Médecins Sans Frontières-OCG
Record Dates: First submitted 2014-02-26; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2013-10

CONDITIONS: Malnutrition
Keywords: malnutrition; children's health; prevention; ready-to-use supplementary food; lipid based nutrient supplement; chad; children
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12 months RUSF (Experimental): Children between 6 to 24 months received ready-to-used supplementary food every months during the whole year.
  Interventions: Dietary Supplement: Ready-to-Used Supplement Food administration
- 4 months RUSF (Active Comparator): children between 6 to 24 months of one zone received a ready-to-used supplement food during the 4 months of the hunger gap period (june to september)
  Interventions: Dietary Supplement: Ready-to-Used Supplement Food administration

INTERVENTIONS:
Dietary Supplement: Ready-to-Used Supplement Food administration
  Other Names: Plumpy 'doz

SUMMARY:
The hypothesis for the study is that 12 months of a Ready-To-Use Supplementary Food (RUSF) distributions have a greater impact on children's health than the standard RUSF distributions during the hunger gap period (june to september). We estimated that the 12 month RUSF will decrease the incidence of severe acute malnutrition by 33% compared to an administration only during the hunger gap period (4 month a year).

ELIGIBILITY:
Inclusion Criteria:

* children between 6 months and 24 months of age

Exclusion Criteria:

* children who can 't swallow
* children from parents who does not want to be in the study

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5700 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of acute severe malnutrition | overall study time, 22 months
  Incidence of acute severe malnutrition will be assessed for the overall 2 years.
  Estimation if incidence will include children from their entry in the study to their exit of study (disharge as 24 months, dead of Lost of follow up )
Mortality rate | overall study time 22 months
  Mortality will be assessed for the overall 2 years. Estimation will include children from their entry in the study to their exit of study (disharge as 24 months, dead of Lost of follow up )

SECONDARY OUTCOMES:
Morbidity | overall study time 22 months
Gain of mid-upper-arm circumference (MUAC) gain | 22 months
Weight for Height gain | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Antierens, Study Chair — Medecins Sans Frontieres, Netherlands; France Broillet, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (1):
- Médecins Sans Frontières-OCG, Massakory, Chad